CLINICAL TRIAL: NCT00131989
Title: Phase I Dose Escalation Trial of the Raf Kinase Inhibitor BAY 43-9006 (NSC #724772) as Single Agent for Adults With Relapsed and Refractory Acute Leukemias and Chronic Myeloid Leukemia in Blast Crisis
Brief Title: Sorafenib in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03154; J-0509; U01CA070095 (NIH)
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-14 or 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a CR may be considered for retreatment with sorafenib for up to an additional 6 courses upon disease recurrence provided the duration of CR is longer than 1 month.
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of sorafenib in treating patients with relapsed or refractory acute myeloid leukemia, acute lymphoblastic leukemia, or chronic myelogenous leukemia. Sorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose-limiting toxicity(s) (DLTs) and maximally tolerated dose (MTD) of BAY 43-9006 given orally.

SECONDARY OBJECTIVES:

I. To obtain preliminary evidence of tumor response to BAY 43-9006 in patients. II. To assess the pharmacokinetic profile of BAY 43-9006. III. To characterize the preliminary profile of adverse events and changes in laboratory parameters in patients treated with BAY 43-9006.

IV. To assess effects of BAY 43-9006 on various cellular properties of leukemic blasts exposed to drug in vivo and in vitro.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive oral sorafenib twice daily on days 1-14 or 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete remission (CR) may be considered for retreatment with sorafenib for up to an additional 6 courses upon disease recurrence provided the duration of CR is longer than 1 month.

Cohorts of 3-6 patients receive escalating doses of sorafenib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 12 patients are treated at the MTD.

After completion of study treatment, patients are followed monthly for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathological confirmation (histologically or cytologically) of relapsed or refractory acute myeloid leukemia (other than acute promyelocytic leukemia), acute lymphocytic leukemia, or chronic myeloid leukemia in blast crisis
* The morphologic diagnosis of AML (non-APL), ALL, and CML in blast crisis will be made independently by members of the hematologic pathology division; routine staining and standard criteria as outlined by the Report of the NCI-Sponsored Workshop will be followed
* All patients must have been refractory to or relapsed from their most recent therapy AND are considered ineligible for potential curative approaches including allogeneic stem cell transplant; in addition, patients must be at least:

  * 3 weeks from last cytotoxic chemotherapy (excluding hydroxyurea)
  * Hydroxyurea may be used for blast count control but must be discontinued within 48 hours of the initiation of BAY 43-9006
  * 2 weeks from last radiation therapy
  * 3 week from last biologic therapy (including myeloid growth factors)
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 2 months
* Multilineage bone marrow failure due to the subject's underlying leukemia
* Total blast count in the peripheral blood < 30,000
* Total bilirubin =< 2 mg/dl
* AST(SGOT)/ALT(SGPT) =< 5 X institutional upper limit of normal
* Serum creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* All women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; the effects of BAY 43-9006 on the developing human fetus at the recommended therapeutic dose are unknown; however, kinase inhibitors are known to be teratogenic; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with APL are not eligible for this clinical trial
* Patients who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Patients with rapidly increasing peripheral blood blast counts (increase in the absolute peripheral blast count > 50% within one week) or uncontrolled (absolute blast count > 30,000) while on hydroxyurea will be excluded
* Patients with uncontrolled hypertension (i.e., persistent grade 3 while undergoing treatment)
* Patients may not be actively receiving any other investigational agents
* Patients active and / or untreated CNS leukemia will not be eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 43-9006
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with BAY 43-9006
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BAY 43-9006; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have any evidence of bleeding diathesis
* Patients must not be on therapeutic anticoagulation; prophylactic anticoagulation (i.e. low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for PT, INR or PTT are met
* Patients must not be taking the cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine, or phenobarbital), rifampin or St. John's wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
DLT defined as non-hematologic > grade 3 or hematologic grade 4 marrow aplasia > 28 days (without leukemia clearance) as assessed by NCI-CTC version 3.0 | 28 days
  Observed toxicities will be reported and summarized s with frequencies, type and grade in a descriptive manner. No formal statistical inference will be made on this dose-finding study.
MDT based on the incidence of DTL as assessed by NCI-CTC version 3.0 | 28 days
  Observed toxicities will be reported and summarized s with frequencies, type and grade in a descriptive manner. No formal statistical inference will be made on this dose-finding study.

SECONDARY OUTCOMES:
Response (CR and/or PR) | Up to 1 year
  Summarized in different dose levels and durations. The 95% confidence intervals will be provided.
Pharmacokinetic parameters | At baseline, at 0.25, 0.5, 1, 2, 4, 6, 8, 24, and 48 hours (days 1, 2, and 3) at days 8, 15, and 29
  Pharmacokinetic parameters over time in different dose levels will be evaluated via descriptive statistics.
Sorafenib tosylate related adverse events as assessed by NCI-CTC version 3.0 | Up to 1 year after completion of treatment
  Adverse events will be summarized with frequencies by type and grade in different dose levels and durations using descriptive statistics.
Impact of sorafenib tosylate on the Raf kinase/MEK/ERK signaling pathway | At baseline and at 28 days (course 1)
  Mean percentage changes will be estimated along with 95% confidence intervals. Dichotomous outcome (on/off) will be tabulated and proportions of activation between pre and post treatment will be compared using Fisher's exact test for each of those targets involved in Raf kinase signaling pathway.

CONTACTS AND LOCATIONS:
Overall Officials: B. Smith, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States